CLINICAL TRIAL: NCT04913649
Title: Intravenous Iron to Treat Postoperative Anemia in Older Cardiac Surgery Patients: a Randomized Controlled Trial'
Brief Title: Intravenous Iron to Treat Postoperative Anemia in Older Cardiac Surgery Patients
Acronym: AGE-ANEMIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: dr. P. Noordzij (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor-Investigator, dr. P. Noordzij, Principal investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL77442.100.21
Record Dates: First submitted 2021-05-28; First posted 2021-06-04 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Iron Deficiency Anemia
Keywords: Cardiac surgery; Postoperative anemia; Intravenous iron; Postoperative disability
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric derisomaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two center randomized controlled trial. Patients will either receive IVI (Monofer) or placebo. Via a computer generated randomization patients will be randomly assigned (1:1) to either a single dose of intravenous ferric derisomaltose (Monofer) 100 mg/mL solution for infusion (intervention group) or intravenous NaCl 0.9% (placebo group) (randomisation with block size 4). Stratification takes surgical intervention (AVR or CABG) and hospital location into account.
Who Masked: Participant, Investigator
Masking Description: Investigator and patient will be blinded for treatment allocation. As the IVI solution is brown and the placebo solution is colourless, the infusion bags and lines will be light-protected in order to prevent identification of the investigational product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous iron (ferric derisomaltose) (Experimental): The intervention consists of a single dose of ferric derisomaltose (Monofer®) 100 mg/mL solution for infusion (Monofer® is a registered product with a marketing authorization in the Netherlands (RVG number: 103070). Manufacturer: Pharmacosmos A/S, Denmark. Dutch marketing authorization holder: Cablon Medical B.V). The method of administration and dosage of the investigational medication are standard treatment. The ferric derisomaltose dose will calculated for each patient depending on body weight (20mg/kg) and diluted in 250 ml NaCl 0.9%. Treatment takes approximately 60 minutes. Vital signs of the patient will be monitored during administration of the investigational medication and for 30 minutes afterwards
  Interventions: Drug: Ferric Derisomaltose 100 MG/ML
- Placebo (Placebo Comparator): Single dose of sodium chloride 0.9% (250ml). Treatment takes approximately 60 minutes. Vital signs of the patient will be monitored during administration of the investigational medication and for 30 minutes afterwards
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Ferric Derisomaltose 100 MG/ML — Postoperative treatment with a single dose IVI (ferric derisomaltose), with a dose of 20mg/kg in approximately 60 minutes.
  Other Names: Monofer
  Arms: Intravenous iron (ferric derisomaltose)
Drug: Sodium chloride — Postoperative treatment with a single dose NaCl 0.9% in approximately 60 minutes.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Postoperative anemia is common in cardiac surgery with cardiopulmonary bypass. Iron deficiency delays the recovery from postoperative anemia and may negatively affect the postoperative trajectory of cardiac surgery patients. The objective of the study is to determine the effect of treatment of postoperative iron deficiency anemia with intravenous iron on disability 90 days after surgery. This will be evaluated in a randomized placebo-controlled double blind two-center trial in which 310 elective cardiac surgery patients will be included.

DETAILED DESCRIPTION:
Rationale: Postoperative anemia is common in cardiac surgery with cardiopulmonary bypass. Iron deficiency delays the recovery from postoperative anemia and may negatively affect the postoperative trajectory of cardiac surgery patients.

Objective: To determine the effect of treatment of postoperative iron deficiency anemia (IDA) with intravenous iron (IVI) on disability 90 days after surgery.

Study design: Randomized placebo-controlled double blind two-center trial

Study population: 310 elderly patients (≥70 years) with moderate postoperative IDA on postoperative day (POD) 1 (hemoglobin (Hb) 85 - 110 g/L, ferritin concentration < 100 µg/L or iron saturation <20%) after uncomplicated elective cardiac surgery (aortic valve repair (AVR) and coronary artery bypass graft (CABG) surgery).

Intervention: Postoperative treatment with a single dose IVI (ferric derisomaltose, Monofer®, N = 155) compared to postoperative treatment with sodium chloride (NaCL) 0.9% (placebo, N = 155).

Main study endpoints: Primary endpoint is disability as measured by the 12- item World Health Organization Disability Assessment score 2.0 (WHODAS-12 at POD 90 after elective cardiac surgery. Secondary endpoints are change in patient reported outcome measures (PROMs) related to dyspnea (assessed with the Rose Dyspnea Score (RDS)) and to health-related quality of life (HRQL) (assessed with The Older Persons and Informal Caregivers-Short Form (TOPICS-SF) questionnaire) at POD 90, the number of postoperative red blood cell (RBC) transfusions, change in reticulocyte hemoglobin content (pg) from randomization to hospital discharge, Hb levels at discharge, hospital complications and days alive and out of hospital at 90 days. Lastly, the difference in functional outcomes (e.g. steep ramp or 6-minute walk test) and Hb value at POD 90 will be assessed as an exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent with age ≥ 70 years
* Elective AVR or CABG surgery
* Expected uncomplicated postoperative trajectory, defined as:
* No inotropic agents or ventilation at time of final inclusion (POD 1)
* Expected discharge to general ward at POD 1
* Moderate postoperative IDA, defined as:
* Hb between 85 and 110 g/L and
* Ferritin <100 µg/L or
* Iron saturation (TSAT) < 20%

Exclusion Criteria:

* Medical history of iron overload/haemochromatosis
* Medical history of liver cirrhosis or ALT/AST value in blood serum triple of normal value (female patients: ALT >120, AST >105 U/L. Male patients: ALT>150, AST>135 U/L)
* Severe renal failure (eGFR<15ml/min/1.73m2)
* Recent treatment with IVI (<12 weeks prior)
* Serious or severe allergic reaction to IVI in medical history
* Severe asthma or eczema in medical history (atopic constitution)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability | 90 days after elective cardiac surgery
  Disability measured by the 12- item World Health Organization Disability Assessment score 2.0 (WHODAS-12). Based on the answers a disability score can be calculated. 0% is no disability and 100% is fully disabled.

SECONDARY OUTCOMES:
Change in patient reported outcome measures (PROMs) related to dyspnea | 90 days after elective cardiac surgery
  PROMS related to dyspnea are assessed with the Rose Dyspnea Scale (RDS). Rose Dyspnea Scale scores range from 0 to 4 with higher scores indicating more dyspnea with common activities.
Change in patient reported outcome measures (PROMs) related to health related quality of life (HRQL) | 90 days after elective cardiac surgery
  HRQL is assessed with The Older Persons and Informal Caregivers-Short Form (TOPICS-SF) questionnaire. The TOPIC-SF is comprised of 22 items in 7 domains of health and well-being. Scores in the different domains ranges from 0 to 5, higher scores indicating diminished quality of life.
Red blood cell transfusions | +/- 7 days after elective cardiac surgery
  Number of red blood cell transfusions during hospital stay
Change in reticulocyte hemoglobin content | +/- 7 days after elective cardiac surgery
  Change in reticulocyte hemoglobin content from randomization to hospital discharge
Change in Hb level | +/- 7 days after elective cardiac surgery
  Change in Hb level from randomization to hospital discharge
Postoperative complications | +/- 7 days after elective cardiac surgery
  Postoperative complications during hospital stay
Days alive and out of hospital | 90 days after elective cardiac surgery
  Days alive and out of hospital

OTHER OUTCOMES:
Functional outcome (exploratory endpoint) | +/- 90 days after elective cardiac surgery
  As part of routine care, patients are offered a cardiac revalidation program supervised by a physical therapist after hospital discharge (POD 90). To assess whether patients can safely start exercising, a functional test is performed (e.g. steep ramp or 6-minute walk test). For this study, the results of these tests will be requested to assess functional capacity after surgery
Change in Hb level at 90 days (exploratory endpoint) | +/- 90 days after elective cardiac surgery
  Laboratory results (i.e. Hb values if available) assessed by the treating cardiologist are requested when patients have visited the hospital during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Peter Noordzij, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Amphia Hospital, Breda
  - St Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smoor RM, Rettig TCD, Vernooij LM, Groenewegen EM, van Dongen HPA, Noordzij PG. The effect of postoperative intravenous iron in anaemic, older cardiac surgery patients on disability-free survival (AGE ANEMIA study): study protocol for a multi-centre, double-blind, randomized, placebo-controlled trial. Trials. 2023 Oct 26;24(1):693. doi: 10.1186/s13063-023-07725-y. PMID 37885026